CLINICAL TRIAL: NCT05650736
Title: JAK1 Inhibition in Granuloma Annulare: an Opportunity for Pathogenesis Directed Therapy
Brief Title: Janus Kinase Inhibition in Granuloma Annulare
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: William Damsky (Other)
Collaborators: Yale University (Other); Pfizer (Industry)
Responsible Party: Sponsor-Investigator, William Damsky, Assistant Professor in Dermatology and Dermatopathology, Yale University
Organization: Yale University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000033312; No NIH funding (Other: 10.11.23)
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-09

CONDITIONS: Granuloma Annulare
Keywords: Granuloma Annulare; Inhibition
MeSH Terms: conditions — Granuloma Annulare; Inhibition, Psychological | interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: moderate to severe GA affecting at least 5% body surface area
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abrocitinib 200 mg daily (Experimental): 6 months of treatment with abrocitinib 200 mg daily
  Interventions: Drug: Abrocitinib 200 mg

INTERVENTIONS:
Drug: Abrocitinib 200 mg — Abrocitinib (Cibinqo) is FDA approved at 200 mg dose once daily for the treatment of atopic dermatitis. It is not currently FDA approved for the treatment of GA.

SUMMARY:
The primary objective is to determine if JAK1 specific inhibition is effective in treating granuloma annulare (GA), a problematic inflammatory skin disease without an FDA approved treatment. The primary outcome will be the percentage change in the body surface area (BSA) involvement by GA after 6 months of treatment with abrocitinib 200 mg daily in 10 patients with moderate to severe GA affecting at least 5% body surface area (BSA).

DETAILED DESCRIPTION:
There are no effective treatments for GA. Systemic corticosteroids can be effective in temporarily controlling GA; however, GA patients are almost never treated with systemic steroids due to the myriad potential adverse effects of this drug class and its transient effect on disease control. Intralesional (intradermal) steroid injections can be effective in patients with localized GA but are not really an option for patients with BSA > 1-2%, require frequent clinic visits for injection, are painful, and also only transiently control disease. A variety of other treatment approaches have been described and include: antibiotics (minocycline, doxycycline, others), hydroxychloroquine, phototherapy, tumor necrosis factor inhibitors, among others. However, these therapies are rarely effective. GA is notoriously recalcitrant to treatment.

With no FDA approved therapies for GA and current approaches being broadly ineffective; there is a large unmet need for an effective treatment. Likely in part because of under recognition, GA is designated as a rare disease by the National Organization for Rare Disorders. Progress in the treatment of GA has been impaired by a poor understanding of disease pathogenesis. Not only will this study allow for greater clarity regarding the pathogenesis of GA, but an oral treatment option for patients that is easier to administer compared to other therapies (such as injections) and with less potential systemic side effects.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Male and female patients 18 years old or older
* Diagnosis of GA with supportive skin biopsy
* BSA involvement of at least 5%
* If patients are on systemic therapies or phototherapy for their GA, they must discontinue these therapies with a washout period of 4 weeks and must remain off them during the study
* If patients are on topical therapies for their GA, they must discontinue these therapies with a washout period of 2 weeks and must remain off them during the study
* Females of childbearing potential must agree to use birth control during the study and there must be a negative pregnancy test documented prior to starting the medication.
* Patients must be willing to have skin biopsies, blood collection, and total body photography and to comply with clinic visits

Exclusion Criteria:

* Age <18 years old
* Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin)
* Patients known to be HIV or hepatitis B or C positive, or have an active, serious infection herpes simplex, herpes zoster, and pneumonia. This would also include localized infections.
* Patients with positive tuberculin skin test or positive QuantiFERON® Tuberculosis test
* Patients with significant hepatic impairment
* Patients with moderate renal impairment
* Patients with uncontrolled peptic ulcer disease
* Patients with a history of deep vein thrombosis and/or pulmonary embolism and/or clotting disorder
* Patients with any history of myocardial infarction or stroke.
* Patients taking concomitant immunosuppressive medications, with the exception of methotrexate and/or low-dose prednisone, including but not limited to mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNF-α inhibitors
* Women of childbearing potential who are unable or unwilling to use birth control while taking the medication
* Women who are pregnant or nursing
* Current smoker or history of any tobacco use
* Screening labs outside the normal range for parameters associated with potential risk for treatment under investigation. Including but not limited to:

  i. Platelets <150,000/mm3 ii. Absolute neutrophil count <1,000/mm3 iii. Hemoglobin levels <8 g/dL iv. Absolute lymphocyte count <500/mm3
* Patients who are taking moderate to strong inhibitors of both CYP2C19 and CYP2C9, or strong CYP2C19 or CYP2C9 inducers, as well as P-gp substrate where small concentration changes may lead to serious or life-threatening toxicities.
* Patients who have received a live vaccine. Patients should wait a minimum of 2 weeks, if recently vaccinated, prior to initiating treatment and should not receive a live vaccine during treatment or 2 weeks post-treatment.
* Patients with any medical, psychiatric, or social condition that is likely to unfavorably affect the risk-benefit of continued study participation, interfere with study compliance or confound safety or efficacy assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in BSA involvement by active GA | Baseline and 6 months
  The percentage change in the body surface area (BSA) involvement by GA after 6 months of treatment with abrocitinib 200 mg daily in 10 patients with moderate to severe GA affecting at least 5% body surface area (BSA).

SECONDARY OUTCOMES:
Changes in Granuloma Annulare Severity and Morphology Instrument (GASMI) score | Baseline and 6 months
  Changes in GASMI score baseline vs. after 6 months of treatment. The Granuloma Annulare Severity and Morphology Instrument is a clinical severity scoring tool for GA. The score is determined by the study team who will examine the participants skin to determine the severity of the GA in different anatomic areas. Scores range from 0-165 with higher score indicating a worse outcome.
Changes in Skindex-16 (Skin related quality of life index) | Baseline and 6 months
  Changes in Skindex-16 (Skin related quality of life index) baseline vs. after 6 months of treatment. This is a 16 item validated skin related Quality of Life questionnaire which will be administered by the study team to assess how GA affects the participants quality of life. Scores range from 0-96, higher scores indicating more significant impact on quality of life.
Changes in molecular signatures in skin and blood before and after treatment | Baseline and 6 months
  Changes in molecular signatures in skin and blood at baseline vs. after 6 months of treatment. Molecular signatures will be assessed in the skin and in the blood. RNA-sequencing will be used to examine transcriptional profiles in this skin. A high throughput proteomic assay will be used to examine molecular profiles in the blood.

CONTACTS AND LOCATIONS:
Overall Officials: William Damsky, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No